CLINICAL TRIAL: NCT04928079
Title: 6-year Follow-up of Dysphagia in Patients With Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: （2020）LunShenYan（ 191 ）
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Dysphagia
Keywords: Parkinson's Disease; dysphagia
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: deep brain stimulation — performing deep brain stimulation if needed
  Other Names: DBS
Drug: Anti-Parkinsonian Drugs — Using anti-parkinsonian drugs if needed
  Other Names: Anti-Parkinsonian medicine

SUMMARY:
We recruited 116 patients with idiopathic PD who were from the Neurology clinic of the Second Affiliated Hospital of Zhejiang University, School of Medicine from January 2014 to November 2014. Perform videofluroscopic swallowing study and psychiatric and neurological evaluations and followed up after 6 years.

DETAILED DESCRIPTION:
In baseline, 116 patients with idiopathic PD were recruited from the Neurology Clinic of the Second Affiliated Hospital of Zhejiang University School of Medicine according to the United Kingdom PD Society Brain Bank Clinical Diagnostic Criteria. They were admitted from January 2014 to November 2014, and were followed up after 6 years.

Perform psychiatric and neurological evaluations. And use Videofluoroscopic swallowing study (VFSS) to assess the swallowing function of PD patients. Added 200mg of barium sulfate to 286ml water to achieve a concentration of 60%. Add a thickener (Ourdiet Swallow, Ourdiet Biotech Co. Ltd, Guangzhou, China) to prepare juice and pudding viscosities, No thickener was added to the liquid viscosity. The patients were advised to have boluses of 3, 5 and 10 ml of the liquid, juice, pudding viscosities in sequence according to the clinician's instructions under X-ray fluoroscopy. The patients ware sitting or standing, The lateral view of the patients' swallow was recorded by a camera (30 frames per second). The radiologist, the clinician, and the rehabilitation therapist completed this examination. Two person analyzed the video in slow motion and frame - by - frame, and record abnormal results. The VFSS inspection parameters are Penetration/aspiration score and Residue score. In order to reduce the influence of drugs on dysphagia, all patients were in the off - period. The patients stopped taking anti-Parkinson's disease drugs from 9 o'clock the night before the examination, and were tested in the morning (free of medicine for more than 12 hours).

The patients had completed the above tests in 2014 and were asked to perform the above assessments again.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD according to the United Kingdom PD Society Brain Bank Clinical Diagnostic Criteria.

Exclusion Criteria:

* (1) Parkinsonian syndromes;(2) with severe lung disease, severe liver insufficiency and cardiac insufficiency; (3) Kubota water drinking test grade ≥3; (4) have had or combined other diseases that affect swallowing function; (5) Nasal feeding, gastric reflux or gastrostomy; (6) Mental disorders Or patients with low intelligence and cognitive function, unable to understand and cooperate with the examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 116 idiopathic PD
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
penetration - aspiration score | in the morning, before taking anti-parkinson drugs
  according to the 8-Point Penetration-Aspiration Scale, PAS ≥ 6 means that material enters below the vocal cords.
residue score | in the morning, before taking anti-parkinson drugs
  evaluate the residue in the oral cavity and pharynx (vallecula, pyriform sinuses) after the first swallowing. Residue amount was rated on a scale from 0 to 3: no residue visible, 0 score; mild residue (less than 25% of the level of the height of the structure), 1 score; moderate residue (25% to 50% of the height of the structure), 2 score; severe residue (high than 50% of the structure height), 3 score.

SECONDARY OUTCOMES:
water swallow test | in the morning, before taking anti-parkinson drugs
  The patient is asked to sit in a chair, and is handed a cup containing 30 mL of water at normal temperature. The patient is then asked to "Please drink this water as you usually do." Time to empty a cup is measured, and the drinking proﬁle and episodes are monitored and assessed.
SDQ-C | in the morning, before taking anti-parkinson drugs
  The Chinese version of the Swallowing Disturbance Questionnaire

OTHER OUTCOMES:
MMSE | in the morning, before taking anti-parkinson drugs
  Mini-mental State Examination (MMSE)；
HAMD | in the morning, before taking anti-parkinson drugs
  Hamilton Depression Scale
HAMA | in the morning, before taking anti-parkinson drugs
  Hamilton Anxiety Scale
H&Y | in the morning, before taking anti-parkinson drugs
  Hoehn-Yahr stage
PDQ-39 | in the morning, before taking anti-parkinson drugs
  Parkinson Disease Quality of Life Measure
NMSQ | in the morning, before taking anti-parkinson drugs
  Non-Motor Symptoms Quest

CONTACTS AND LOCATIONS:
Overall Officials: Wei Luo, PhD, Principal Investigator — the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Result] Argolo N, Sampaio M, Pinho P, Melo A, Nobrega AC. Videofluoroscopic Predictors of Penetration-Aspiration in Parkinson's Disease Patients. Dysphagia. 2015 Dec;30(6):751-8. doi: 10.1007/s00455-015-9653-y. Epub 2015 Oct 22. PMID 26492880
- [Result] Fukuoka T, Ono T, Hori K, Wada Y, Uchiyama Y, Kasama S, Yoshikawa H, Domen K. Tongue Pressure Measurement and Videofluoroscopic Study of Swallowing in Patients with Parkinson's Disease. Dysphagia. 2019 Feb;34(1):80-88. doi: 10.1007/s00455-018-9916-5. Epub 2018 Jun 8. PMID 29948261